CLINICAL TRIAL: NCT04962048
Title: The Influence of Pulse-synchronized Negative Pressure on the Dermal Microcirculation
Acronym: PSyNeP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results not goal-oriented, premature termination.
Sponsor: Orputec (Other)
Collaborators: Medical University of Graz (Other); Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSyNeP
Record Dates: First submitted 2021-06-17; First posted 2021-07-14 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Microcirculation; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: After ensuring a comfortable position, each subject will receive treatment with the pulse-synchronized negative pressure (PSNP) device on one randomly chosen lower leg for 120 minutes.The non-invasive imaging (Laser-Doppler Imaging = LD , Hyperspectral Imaging = HS, Thermal Imaging = TH) will be performed before and after the intervention.
  This treatment course will be applied twice a day (with 4h +/- 2h in between) for two consecutive days. Toleration of the treatment and wellbeing of the subjects will be assessed by a Visual Analogue Scale.
  Finally, another series of imaging (LD, HS, TH) will be performed on the morning of the third day without a prior intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulse-synchronized negative pressure (PSNP) device (Experimental): One leg will be treated with the pulse-synchronized negative pressure (PSNP). The other leg serves as non-treated control.
  Interventions: Device: pulse-synchronized negative pressure (PSNP) device; Other: Control - no intervention

INTERVENTIONS:
Device: pulse-synchronized negative pressure (PSNP) device — The machine consists of four components: an electrocardiograph (ECG), a vacuum pump, a software computing the timing of suction and drainage, and an individual suction cap for each patient. One leg will be treated with the PSNP-device. The treatment course with PSNP will be applied twice a day (with 4h +/- 2h in between) for two consecutive days.
Other: Control - no intervention — The other leg serves as non-treated control

SUMMARY:
The technology of the pulse-synchronous alternating pressure system has been patented and is ready for application. Since the device is a combination of commercially available products with a software controlling the duration/initiation of the negative pressure, no harm for the study participant is expected. With no adequate preclinical model of impaired microcirculation being available, and due to the non-invasive nature of the device, the rationale to test the product in a controlled setting in clinical patients is justified. The intervention takes place twice a day for two consecutive days with objective assessment of the microcirculation before and after the intervention. Thereby, the immediate effect of the intervention is to be evaluated. A fifth assessment takes place on the third day without prior intervention to assess a possible long-term effect (comparison against first measurement - base line).

The primary aim of this project is to investigate the tolerability and the comfort of pulse-synchronized negative pressure (PSNP) applied by the device manufactured by Orputec GmbH on the dermal microcirculation. Evaluation of patient comfort and tolerability will be performed by a Numerical Rating Scale (NRS).

The application of the device (PSNP) significantly influences the dermal microcirculation (measuring by LD, HS, TH).

The aims of this project is to investigate the tolerability / comfort and the effect of pulse-synchronized negative pressure (PSNP) applied by the device manufactured by Orputec GmbH on the dermal microcirculation. Objective evaluation of microcirculation with laser doppler (LD), hyperspectral imaging (HS), thermal imaging (TH).

DETAILED DESCRIPTION:
Orputec has developed a device that uses the technology of a pulse-synchronized alternating pressure system. It can be applied in the field of regenerative medicine to treat lymphedema by improving the blood- and lymphatic circulation. The machine consists of four components: an electrocardiograph (ECG), a vacuum pump, a software controlling the timing of suction and drainage, and an individual suction cap for each patient.

The study is designed as an open, interventional cohort, intraindividually controlled, pilot study. A pilot sample size of 12 is chosen because the device will be tested in a controlled setting for the first time. No formal sample size calculation was performed.

The collective consists of 12 subjects, with diabetes mellitus (DM) type 2 but no apparent wounds on the lower leg. Before inclusion, subjects will be screened for current skin lesions in the region of interest (ROI), comorbidities, and their medical history concerning diabetes and skin lesions. The ROI on both lower legs will be marked, and the dermal microcirculation will be measured, non-invasively, using LD, HS, and TH. After ensuring a comfortable position, each subject will receive treatment with the PSNP device on one chosen lower leg for 120 minutes. During the treatment, a warming unit, which is also used after flap surgery to maintain an adequate ambient temperature, will be used to obtain local thermal hyperaemia, hence a prospected dilation of the vessels. The non-invasive imaging (LD, HS, TH) will be performed before and after the intervention. This treatment course will be applied twice a day (with 4h +/- 2h in between) for two consecutive days. Toleration of the treatment and wellbeing of the subjects will be assessed by a Visual Analog Scale (VAS). Finally, another series of imaging (LD, HS, TH) will be performed on the morning of the third day without a prior intervention.

Statistical analysis of numeric endpoints: All numeric endpoints will be checked for normality, e.g. by using a Shapiro-Wilk test. If a numeric endpoint deviates from normality, then data transformations (e.g. log-transformation) will be considered. Numeric endpoints will be analysed by means of a repeated measures analysis of variance (ANOVA). The level of significance will be set to 5% in all analyses. No adjustment for multiple comparisons will be performed.

Additionally, the following comparisons will be performed by using descriptive statistics (e.g. Q1, median, Q3, mean, standard deviation) and graphical methods (e.g. box plots):

* Comparison of time points (prior to intervention on day 1; after intervention on day 1; prior to control on day 1; after control on day 1 and day 3) within each treatment condition (intervention: treated leg; control: untreated leg).
* Comparison of treatment conditions (treated vs. untreated legs) for each time point.

In order to identify influencing factors for the effect of the PSNP treatment, the investigators will use graphical methods as well as regression models and mixed effects models (e.g., analysis of covariance).

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals suffering from DM type 2 and willing to participate in this study
* First diagnosis of DM type 2 at least 10 years prior to inclusion OR presence of diabetic dermopathy.
* Age: 45-99
* Written consent of the participant after being informed

Exclusion Criteria:

* Skin lesions or dermatoses in the region of interest (ROI)
* Non-ability to comprehend the nature and course of the study

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change of toleration / wellbeeing due to intervention of PSNP with Numeric Rating Scale | 2 times on day 1 and day 2
  Successful intervention with the PSNP device without harm to the patients. Change of toleration of the treatment and wellbeing of the subjects will be assessed by a Numerical Rating Scale (scale 0 - 10)

SECONDARY OUTCOMES:
Change of microcirculation with laser doppler (LD) | 4 times on day 1 and 2; once on day 3
  LD is measuring the blood flow: Blood flow is then calculated in a unit called Flux based on the red cell concentration in red cell velocity. The blood flow correlates directly to the microcirculation in the skin. A higher blood flow indicates a better microcirculation.
Change of microcirculation with hyperspectral imaging (HS) | 4 times on day 1 and 2; once on day 3
  HS is measuring oxygenation in the blood: The oxygenation index is given in percent. The oxygenation correlates directly to the microcirculation in the skin. A higher blood oxygenation indicates a better microcirculation.
Change of microcirculation with thermal imaging (TH) | 4 times on day 1 and 2; once on day 3
  Objective evaluation of microcirculation with thermal imaging (TH). TH is measuring the skin temperature in Kelvin. The skin temperature correlates directly to the blood flow and the microcirculation in the skin. A higher skin temperature indicates a better microcirculation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Peter Kamolz, Univ.-Prof., Principal Investigator — Medical University of Graz, Graz, Styria, Austria
Locations (1):
- Division of Plastic, Aesthetic and Reconstructive Surgery, Graz, Styira, Austria